CLINICAL TRIAL: NCT05095467
Title: Prospective Study With HIPEC-AS in Patients With Locally Advanced, Limited or Extensive Peritoneal Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Brief Title: HIPEC-AS in Patients With Peritoneal Metastasis of the Stomach or Esophagogastric Junction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xuefei.Wang (Other)
Responsible Party: Sponsor-Investigator, Xuefei.Wang, Professor, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2021-574
Record Dates: First submitted 2021-10-25; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Stomach Neoplasms; Peritoneal Metastases
Keywords: Stomach Neoplasms; Peritoneal Metastases; Hyperthermic Intraperitoneal Chemotherapy; paclitaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): patients with locally resectable GC (cT4aNxM0, P0)
  1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), surgery+HIPEC, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3)
  Interventions: Procedure: HIPEC; Drug: Paclitaxel-albumin; Drug: Tegafur-gimeracil-oteracil potassium; Procedure: Surgery+HIPEC
- Group B (Experimental): patients with peritoneal metastasis stage P1a or P1b (cTxNxM1, P1a or P1b)
  1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), surgery+HIPEC, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3)
  Interventions: Procedure: HIPEC; Drug: Paclitaxel-albumin; Drug: Tegafur-gimeracil-oteracil potassium; Procedure: Surgery+HIPEC
- Group C (Experimental): group C is patients with peritoneal metastasis stage P1c (cTxNxM1, P1c)
  1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3)
  Interventions: Procedure: HIPEC; Drug: Paclitaxel-albumin; Drug: Tegafur-gimeracil-oteracil potassium

INTERVENTIONS:
Procedure: HIPEC — The abdominal cavity will be filled with paclitaxel 120mg/m2 heated at 43℃ for 1 hour with a hyperthermic circulation machine.
  Other Names: Paclitaxel injection
Drug: Paclitaxel-albumin — albumin paclitaxel D1, D8; S-1: D1-D14
Drug: Tegafur-gimeracil-oteracil potassium — 40mg bid(BSA<1.5 m2) ，60mg bid(BSA>=1.5 m2); D1-D14, po, bid.
Procedure: Surgery+HIPEC — gastrectomy with D2 lymphadenectomy+HIPEC procedure
  Arms: Group A; Group B

SUMMARY:
HIPEC-AS01 is an open, prospective, single-center phase II clinical study, which will include "cT4aNxM0, P0 or cTxNxM1, P1" patients with gastric or esophagogastric junction adenocarcinoma, to evaluate the efficacy and safety of systemic chemotherapy with HIPEC combined with AS in the perioperative period. Patients enrolled will be divided into three groups. Among them, group A is the patients with locally resectable GC; group B is patients with peritoneal metastasis stage P1a or P1b, group C is patients with peritoneal metastasis stage P1c. The primary purpose is to evaluate the 3-year overall survival rate.

DETAILED DESCRIPTION:
HIPEC-AS01 is an open, prospective, single-center phase II clinical study, which will include Patients With cT4aNxM0, P0, or cTxNxM1*, P1 Adenocarcinoma of the Stomach or Esophagogastric Junction, to evaluate the efficacy and safety of systemic chemotherapy with HIPEC combined with AS in the perioperative period.

Patients enrolled will be divided into three groups. Among them, group A is the patients with locally resectable GC; group B is patients with peritoneal metastasis stage P1a or P1b, group C is patients with peritoneal metastasis stage P1c.

Intervention:

Group A: 1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), surgery+HIPEC, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3).

Group B: 1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), surgery+HIPEC, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3).

Group C: 1 cycle HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy (AS plan, Q21d × 3), HIPEC+S-1 chemotherapy, sequential 3 cycles of chemotherapy ( AS plan, Q21d × 3).

In this study, the patient's overall survival was the main evaluation index. It is estimated that the case recruitment will be completed in 2 years, and the follow-up time will be 3 years. The total sample size is approximately 157 cases.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old ≤ age ≤ 75 years old;
2. The primary gastric lesion was diagnosed as gastric or esophagogastric junction adenocarcinoma (papillary adenocarcinoma, tubular adenocarcinoma, mucinous adenocarcinoma, signet ring cell carcinoma, and poorly differentiated adenocarcinoma. )
3. The tumor is located in the stomach or esophagogastric junction (Siewert type II/III)
4. The preoperative clinical staging is cT4aNxM0, P0 or cTxNxM1*, P1 (*no other distant metastases except peritoneal metastasis)
5. Good bone marrow reserve function: HB≥90g/L; ANC ≥1.5×10*9/L; PLT ≥80×10*9/L
6. Good liver and kidney function reserve: BIL ≤ 1.5 times the upper limit of normal (ULN); ALT and AST ≤ 2.5×ULN; Crea≤1×ULN;
7. Good coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN, activated partial thromboplastin time (APTT) ≤ 1.5 times ULN
8. ECOG (Eastern Cooperative Oncology Group) physical status score 0-2;
9. No prior treatment of chemotherapy, radiotherapy, targeted therapy, immunotherapy, etc;
10. Written informed consent.

Exclusion Criteria:

1. There are distant metastases other than peritoneal metastases;
2. Complications of gastric cancer require emergency treatment, such as bleeding, perforation, obstruction, etc.;
3. Suffer from other malignant tumors within five years;
4. Body temperature ≥38℃ or complicated with infectious diseases requiring systemic treatment;
5. If there is a history of uncontrolled epilepsy, central nervous system disease, or mental disorder, the investigator will determine whether the clinical severity hinders the signing of informed consent or affects the patient's compliance with oral medications;
6. Clinically serious (ie active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) grade II or more severe congestive heart failure, or severe arrhythmia requiring drug intervention, or recent history of myocardial infarction within 12 months;
7. Severe respiratory diseases;
8. Severe liver and kidney dysfunction;
9. Upper gastrointestinal obstruction or abnormal physiological function or malabsorption syndrome, which may affect the absorption of oral drugs;
10. Diseases such as severe diabetes, hyperthyroidism and hypothyroidism have not been clinically controlled.
11. Those who continue to use glucocorticoid therapy within 1 month (except for local application) or who require immunosuppressive therapy for organ transplantation;
12. Pregnant or lactating women;
13. The patient has participated or is participating in other clinical studies (within 6 months);

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
3-year Overall Survival, OS | 3 years
  The time from the date of enrollment of the patient to the date of death or the date of the last follow-up

SECONDARY OUTCOMES:
3-year Progression Free Survival, PFS | 3 years
  The time from the date of enrollment of the patient to the first occurrence of disease progression or death from any cause.
NCI CTC Adverse Events Version 4.0 | 1 year
  Safety of HIPEC-AS plan

CONTACTS AND LOCATIONS:
Overall Officials: Xuefei Wang, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No